CLINICAL TRIAL: NCT02760719
Title: The Effectiveness of Nebulized 3% Hypertonic Saline With Salbutamol in Acute Bronchiolitis in Hospitalised Children- a Randomized Clinical Trial
Brief Title: The Effectiveness of Nebulized Hypertonic Saline Solution for Acute Bronchiolitis
Acronym: NHSAB
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: No relevant data
Sponsor: University Medical Centre Ljubljana (Other)
Responsible Party: Principal Investigator, Tina Plankar Srovin, MD, PhD, University Medical Centre Ljubljana
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22k/12/12
Record Dates: First submitted 2016-04-06; First posted 2016-05-04 (Estimated); Last update posted 2019-08-05 (Actual); Status verified 2019-08

CONDITIONS: Bronchiolitis
Keywords: 3% hypertonic solution; duration of hospitalisation
MeSH Terms: conditions — Bronchiolitis | interventions — Hypertonic Solutions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- hypertonic saline (Experimental): 4 ml of nebulized 3 % hypertonic saline + salbutamol 0,03 ml/kg every 8 hours for the time of hospitalisation and standard supportive care (oxygen to correct hypoxia, minimal handling to minimise the risk of exhaustion, provision of fluids, gentle nasal aspiration)
  Interventions: Drug: nebulized 3% hypertonic solution
- supportive care (No Intervention): Standard supportive care (oxygen to correct hypoxia, minimal handling to minimise the risk of exhaustion, provision of fluids, gentle nasal aspiration)

INTERVENTIONS:
Drug: nebulized 3% hypertonic solution — already described
  Arms: hypertonic saline

SUMMARY:
This study evaluates the effectiveness of nebulized 3% hypertonic saline solution with salbutamol in the treatment of children under 2 years, hospitalised for acute viral bronchiolitis. Half of the participants will receive nebulized 3% hypertonic saline solution with salbutamol three times daily, the other half will receive standard supportive care, which is the cornerstone of the bronchiolitis management.

DETAILED DESCRIPTION:
Acute viral bronchiolitis is the most common lower respiratory tract infection in infants up to two years old. Currently there is no effective treatment so standard treatment remains supportive care with supplemental oxygen to correct hypoxia, minimal handling to minimise the risk of exhaustion and the provision of fluids.

In recent years some studies have suggested that nebulised hypertonic saline, which improve airway hygiene, may influence the course of the illness and reduce the duration of hospitalisation without significant side effects.

Study protocol: half of the included patients will receive standard treatment for bronchiolitis, which includes only supportive care, the other half will additionally receive nebulized 3% hypertonic saline solution with salbutamol (to avoid potential bronchial obstruction) three times daily.

ELIGIBILITY:
Inclusion Criteria:

* first episode of bronchiolitis: viral lower respiratory tract infection with signs of airway obstruction (hyperinflated lungs, tachypnea, increased work of breathing) and crepitations on auscultations
* admission to the hospital
* Wang CSS between 3 and 9
* randomisation within 4 hours of admission

Exclusion Criteria:

* a history or previous episodes of bronchiolitis/bronchitis
* primary diseases: gastro-oesophageal reflux, chronic cardiac or pulmonary diseases including suspected asthma, immunodeficiency, conditions with hypotonia where more severe course of bronchiolitis is expected
* newborns
* premature infants born < 36 weeks of gestation
* oxygen saturation < 85% and patients requiring admission to high dependency or intensive care units at presentation

Ages: 1 Month to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2015-12; Primary Completion 2019-07 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
Fit to discharge time | Outcome measure will be assessed in hours, data will be presented through study completion- estimated to 2 years
  Fit to discharge time: as the point (measured in hours) at which the infant was feeding adequately (taking >75% of their usual intake) and had been in air with a saturation of at least 92% for 6 h.

SECONDARY OUTCOMES:
Duration of hospitalisation | Outcome measure will be assessed in hours, data will be presented through study completion- estimated to 2 years
  Actual time to discharge in hours, which could be prolonged for other reasons than just bronchiolitis
Duration of hypoxia | Outcome measure will be assessed in hours, data will be presented through study completion- estimated to 2 years
  For how long (in hours) participants need the oxygen therapy (have saturation on air bellow 92%).
Clinical severity score (CSS) assessed by Wang score | Through study completion - estimated to 2 years, the patients will be assessed through whole hospitalisation time
  Wang 1992 CSS as an outcome: measured two times daily
Number of participants with treatment related adverse events assessed by questionnaire | Through study completion - estimated to 2 years, the patients will be assessed through whole hospitalisation time
  To asses all possible side effects related to the inhalation of hypertonic saline
Number of participants transferred to the intensive care unit (ICU) | Through study completion - estimated to 2 years, the patients will be assessed through whole hospitalisation time
  The need to be transferred to the ICU because of the respiratory failure
Number of patients readmitted to the hospital because of the same diagnose | Through study completion - estimated to 2 years; the patients will be assessed up to one month after discharge
  Rate of readmission within one month after discharge because of the same disease
Comparison of fit to discharge time between patients treated with nebulized hypertonic saline with respiratory syncytial virus (RSV) versus non-RSV bronchiolitis. | Outcome measure will be assessed in hours, data will be presented through study completion- estimated to 2 years
  To see if there are any differences in fit to discharge time (the point measured in hours at which the infant was feeding adequately - taking >75% of their usual intake and had been in air with a saturation of at least 92% for 6 h) between patients who received nebulized hypertonic saline and have RSV bronchiolitis and patients who received nebulized hypertonic saline and have non-RSV bronchiolitis (to see if hypertonic saline has better effect on fit to discharge time in patients who have RSV bronchiolitis compared to patients who have non-RSV bronchiolitis).
Comparison of hypoxia duration between patients treated with nebulized hypertonic saline with respiratory syncytial virus (RSV) versus non-RSV bronchiolitis. | Outcome measure will be assessed in hours, data will be presented through study completion- estimated to 2 years
  To see if there are any differences in hypoxia (for how long in hours participants need the oxygen therapy: have saturation bellow 92%) between patients who received nebulized hypertonic saline and have RSV bronchiolitis and patients who received nebulized hypertonic saline and have non-RSV bronchiolitis.
Number of participants with treatment related adverse events assessed by questionnaire: comparison of patients with RSV bronchiolitis and patients with non-RSV bronchiolitis. | through study completion - estimated to 2 years, the patients will be assessed through whole hospitalisation time
  To asses all possible side effects related to the inhalation of hypertonic saline in patients who have RSV bronchiolitis compared to the patients who have non-RSV bronchiolitis.

CONTACTS AND LOCATIONS:
Overall Officials: Tatjana Lejko Zupanc, MD, PhD, Study Chair — University Medical Centre Ljubljana
Locations (1):
- Department of infectious disease, University Medical Centre, Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Zhang L, Mendoza-Sassi RA, Wainwright C, Klassen TP. Nebulised hypertonic saline solution for acute bronchiolitis in infants. Cochrane Database Syst Rev. 2013 Jul 31;(7):CD006458. doi: 10.1002/14651858.CD006458.pub3. PMID 23900970
- [Result] Everard ML, Hind D, Ugonna K, Freeman J, Bradburn M, Cooper CL, Cross E, Maguire C, Cantrill H, Alexander J, McNamara PS; SABRE Study Team. SABRE: a multicentre randomised control trial of nebulised hypertonic saline in infants hospitalised with acute bronchiolitis. Thorax. 2014 Dec;69(12):1105-12. doi: 10.1136/thoraxjnl-2014-205953. PMID 25389139
- [Result] Zhang L, Mendoza-Sassi RA, Klassen TP, Wainwright C. Nebulized Hypertonic Saline for Acute Bronchiolitis: A Systematic Review. Pediatrics. 2015 Oct;136(4):687-701. doi: 10.1542/peds.2015-1914. PMID 26416925